CLINICAL TRIAL: NCT00748410
Title: An Open Label, 7-day Repeat Dose Study to Evaluate the Pharmacodynamics of SB-656933-AAA in Patients With Ulcerative Colitis.
Brief Title: Study to Evaluate the Pharmacodynamics of SB-656933 in Patients With Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: SB-656933 is no longer being developed for ulcerative colitis.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUC111342; 2007-005520-32 (EudraCT Number)
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Colitis, Ulcerative
Keywords: CD11b; Ulcerative colitis; 99mTc-HMPAO-labelled leukocyte scintigraphy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — SB 656933

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 7 Days Repeat Dose (Experimental)
  Interventions: Drug: SB-656933

INTERVENTIONS:
Drug: SB-656933 — 7 days repeat dose
  Other Names: SB656933

SUMMARY:
This study will involve the use of a new compound, SB-656933. Accumulation of inflammatory white blood cells (mostly polymorphonuclear neutrophils)in the gut (colon) may be contributing to the pathology of ulcerative colitis. It has been shown that SB-656933 reduces polymorphonuclear neutrophils (PMN) accumulation in pre-clinical models of colitis. 99m-Tc-HMPAO scintigraphy is a imaging technique which will be used in this study to observe the effect of SB656933 on the migration of PMN to inflamed tissue.

ELIGIBILITY:
Inclusion criteria:

* A history of ulcerative colitis for at least 3 months
* moderately active UC, either stable on medications or in a flare of the disease
* Mayo endoscopic score of 2 or 3 within 2 days of dosing.
* Male or female between 18 and 65 years of age
* Women of child bearing potential must use an effective method of contraception.
* Male subjects must agree to use one of the specified contraception method,
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) normal at study start.
* Signed written informed consent
* QTcB or QTcF < 450msec at screening

Exclusion criteria:

* The subject has a positive pre-study drug/alcohol screen.
* A positive test for HIV, hepatitis B or C.
* History of regular alcohol consumption within 6 months of the study
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives prior to the first dose of study medication
* Known allergies
* recent participation in another trial
* recent blood donation
* Pregnant or lactating females
* unwillingness or inability to follow study procedures
* consumption of red wine, seville oranges, grapefruit or grapefruit juice in last 7 seven day before study start.
* Mild UC, Mayo endoscopic score of 0 or 1.
* Toxic megacolon or perforation on plain abdominal Xray.
* Crohn's Disease, indeterminate colitis, bleeding disorders, or active ulcer disease.
* Previous colonic surgery.
* Current or recurrent disease, other than UC, that could affect the action, absorption or disposition of the study medication, or clinical or laboratory assessments.
* Absolute neutrophil count below 2.0x109/L.
* A positive culture for enteric pathogens that is clinically significant, presence of clostridium difficile toxin, or with ova and parasites detected by microscopy, or has a clinical suspicion of an infectious disease of the bowel.
* Symptomatic GI stricture within 6 months of screening or obstructive symptoms within 3 months of screening.
* Likely to require abdominal surgery within the study period.
* Congenital or acquired immunodeficiency, including any immunologic diseases with gastrointestinal involvement except for UC.
* Ongoing neoplastic disease of the bowel.
* History of prostatitis, epididymitis, epididymal cysts, structural abnormalities or testicular cancer.
* Subjects with abnormalities of the renal tract, renal stones or history of recurrent urinary tract infections (UTI.s).
* Subjects with any history of autoimmune hepatitis or sclerosing cholangitis. Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden.
* Blood pressure persistently ≥ 140/90 mmHg at screening
* Concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, renal, pulmonary, hepatic, endocrine, metabolic, haematological, or neurological condition).
* Clinically significant hepatic impairment(Evidence of cirrhosis, Clinical episodes of jaundice)
* Current evidence of, or has been treated for a malignancy within the past 5 years.
* BMI <18 kg.m2 or >35 kg/m2
* Clinically significant renal laboratory values.
* Has not discontinued any prohibited concomitant medication prior to the screening visit or within the protocol-specified time period.
* Has not remained on a stable dose of any permitted concomitant medication(s) for the protocol-specified time period preceding the Screening Visit.
* history of substance abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2009-12-12 (Actual); Study Completion 2009-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3 participants were enrolled and randomized from 22 January 2009 to 12 December 2009. This study was conducted at Academic Medical Centre, Amsterdam, The Netherlands. The study was early terminated on 17 February 2010.
Groups:
- SB656933 20 Milligram (mg): Participants received SB656933 20 mg (10 mg per dose ) tablet administered orally with 240 milliliter(mL) of tepid water on every morning of Day 1 to 7 of the treatment period.
- SB656933 100 mg: Participants received SB656933 100 mg (50 mg per dose ) tablet administered orally with 240 mL of tepid water on every morning of Day 1 to 7 of the treatment period.
Period: Overall Study
Arm/Group | SB656933 20 Milligram (mg) | SB656933 100 mg
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SB656933 20 mg: Participants received SB656933 20 mg (10 mg per dose ) tablet administered orally with 240 mL of tepid water on every morning of Day 1 to 7 of the treatment period.
- Total: Total of all reporting groups
Arm/Group | SB656933 20 mg | SB656933 100 mg | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (0.00) | 39 (15.56) | 46 (15.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 1 and 7 Days Treatment With Daily Dose of SB-656933-AAA in 99m(Technetium-hexamethyl Derivative of Propylene Amine Oxide)Tc-HMPAO Leukocyte Single Photon Emission Computerized Tomography (SPECT) Scintigraphic Activity Scores (SAS)
Description: Data has been presented for participants since change from Baseline data was not analyzed. For scintigraphy, blood was obtained for radiolabelling. Labelled white cells were then injected for SPECT scintigraphy and scanning began 45 minutes after injection of labelled White blood cells (WBCs). SPECT images of the colon were divided into 5 segments: ascending colon, transverse colon, descending colon, sigmoid, and rectum.T he SPECT segment uptake ratio was expressed as a fraction of bone marrow activity obtained from counts in the lumbar spine. The SPECT segment uptake ratio was converted into a four-point (0 to 3) segmental SPECT severity score where grade 0 was equal to no uptake. Only 3 participants were included before the study was discontinued.It was not possible to draw any meaningful conclusions from the very limited data available. Data has been presented for the 3 participants (99001, 99002 and 99003) since the analysis was not done. Baseline was Day -1.
Time Frame: Baseline (Day -1) and Day 1 and 7
Population: The 'All Subjects population' was defined as all participants who received at least one dose of study medication. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Score on scale
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
Score on scale
  99001, Descending colon, Day 1: number analyzed (Participants) | 0 | 1
  99001, Descending colon, Day 1 |  | 1
  99001, Descending colon, Day 7: number analyzed (Participants) | 0 | 1
  99001, Descending colon, Day 7 |  | 1
  99003, Sigmoid, Day 1: number analyzed (Participants) | 0 | 1
  99003, Sigmoid, Day 1 |  | 1
  99003, Sigmoid, Day 7: number analyzed (Participants) | 0 | 1
  99003, Sigmoid, Day 7 |  | 1
  99001, Sigmoid, Day 1: number analyzed (Participants) | 0 | 1
  99001, Sigmoid, Day 1 |  | 2
  99001, Sigmoid, Day 7: number analyzed (Participants) | 0 | 1
  99001, Sigmoid, Day 7 |  | 1
  99002, Rectum, Day 1: number analyzed (Participants) | 1 | 0
  99002, Rectum, Day 1 | 2 |
  99002, Rectum, Day 7: number analyzed (Participants) | 1 | 0
  99002, Rectum, Day 7 | 3 |
  99003, Rectum, Day 1: number analyzed (Participants) | 0 | 1
  99003, Rectum, Day 1 |  | 1
  99003, Rectum, Day 7: number analyzed (Participants) | 0 | 1
  99003, Rectum, Day 7 |  | 1
  99001, Rectum, Day 1: number analyzed (Participants) | 0 | 1
  99001, Rectum, Day 1 |  | 2
  99001, Rectum, Day 7: number analyzed (Participants) | 0 | 1
  99001, Rectum, Day 7 |  | 1

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to follow-up (7 to 10 days after last dose)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
Participants
  Any AE | 1 | 1
  Any SAE | 0 | 0

3. Secondary Outcome: Vital Signs Assessment- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign measurements included SBP and DBP at Day 1 and 7. Data was collected in supine position. It was not possible to draw any meaningful conclusions from the very limited data available. Data has been presented for the 3 participants (99001, 99002 and 99003) since the analysis was not done.
Time Frame: Day 1 and 7
Population: All subject population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: millimeter of mercury (mmHg)
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
millimeter of mercury (mmHg)
  DB: 99001, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 1, pre-dose |  | 90
  DB: 99001, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 1, 1 hour |  | 96
  DB: 99001, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 1, 4 hour |  | 98
  DB: 99001, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 1, 8 hour |  | 83
  DB: 99001, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 7, pre-dose |  | 78
  DB: 99001, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 7, 1 hour |  | 82
  DB: 99001, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 7, 4 hour |  | 89
  DB: 99001, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  DB: 99001, Day 7, 8 hour |  | 99
  SB: 99001, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 1, pre-dose |  | 135
  SB: 99001, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 1, 1 hour |  | 131
  SB: 99001, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 1, 4 hour |  | 138
  SB: 99001, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 1, 8 hour |  | 129
  SB: 99001, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 7, pre-dose |  | 113
  SB: 99001, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 7, 1 hour |  | 120
  SB: 99001, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 7, 4 hour |  | 133
  SB: 99001, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  SB: 99001, Day 7, 8 hour |  | 152
  DB: 99003, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 1, pre-dose |  | 69
  DB: 99003, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 1, 1 hour |  | 63
  DB: 99003, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 1, 4 hour |  | 77
  DB: 99003, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 1, 8 hour |  | 61
  DB: 99003, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 7, pre-dose |  | 55
  DB: 99003, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 7, 1 hour |  | 64
  DB: 99003, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 7, 4 hour |  | 61
  DB: 99003, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  DB: 99003, Day 7, 8 hour |  | 71
  SB: 99003, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 1, pre-dose |  | 108
  SB: 99003, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 1, 1 hour |  | 109
  SB: 99003, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 1, 4 hour |  | 122
  SB: 99003, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 1, 8 hour |  | 106
  SB: 99003, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 7, pre-dose |  | 108
  SB: 99003, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 7, 1 hour |  | 109
  SB: 99003, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 7, 4 hour |  | 110
  SB: 99003, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  SB: 99003, Day 7, 8 hour |  | 123
  DB: 99002, Day 1, pre-dose: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 1, pre-dose | 68 |
  DB: 99002, Day 1, 1 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 1, 1 hour | 63 |
  DB: 99002, Day 1, 4 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 1, 4 hour | 62 |
  DB: 99002, Day 1, 8 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 1, 8 hour | 81 |
  DB: 99002, Day 7, pre-dose: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 7, pre-dose | 59 |
  DB: 99002, Day 7, 1 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 7, 1 hour | 64 |
  DB: 99002, Day 7, 4 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 7, 4 hour | 66 |
  DB: 99002, Day 7, 8 hour: number analyzed (Participants) | 1 | 0
  DB: 99002, Day 7, 8 hour | 72 |
  SB: 99002, Day 1, pre-dose: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 1, pre-dose | 111 |
  SB: 99002, Day 1, 1 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 1, 1 hour | 118 |
  SB: 99002, Day 1, 4 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 1, 4 hour | 110 |
  SB: 99002, Day 1, 8 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 1, 8 hour | 119 |
  SB: 99002, Day 7, pre-dose: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 7, pre-dose | 102 |
  SB: 99002, Day 7, 1 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 7, 1 hour | 99 |
  SB: 99002, Day 7, 4 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 7, 4 hour | 114 |
  SB: 99002, Day 7, 8 hour: number analyzed (Participants) | 1 | 0
  SB: 99002, Day 7, 8 hour | 117 |

4. Secondary Outcome: Vital Signs Assessment- Heart Rate
Description: Vital sign measurements included heart rate at Day 1 and 7. Data was collected in supine position. It was not possible to draw any meaningful conclusions from the very limited data available. Data has been presented for the 3 participants (99001, 99002 and 99003) since the analysis was not done.
Time Frame: Day 1 and 7
Population: All subjects population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: beats per minute (bpm)
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
beats per minute (bpm)
  heart rate: 99001, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 1, pre-dose |  | 85
  heart rate: 99001, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 1, 1 hour |  | 80
  heart rate: 99001, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 1, 4 hour |  | 80
  heart rate: 99001, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 1, 8 hour |  | 77
  heart rate: 99001, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 7, pre-dose |  | 80
  heart rate: 99001, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 7, 1 hour |  | 77
  heart rate: 99001, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 7, 4 hour |  | 80
  heart rate: 99001, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99001, Day 7, 8 hour |  | 87
  heart rate: 99003, Day 1, pre-dose: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 1, pre-dose |  | 60
  heart rate: 99003, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 1, 1 hour |  | 62
  heart rate: 99003, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 1, 4 hour |  | 60
  heart rate: 99003, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 1, 8 hour |  | 71
  heart rate: 99003, Day 7, pre-dose: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 7, pre-dose |  | 73
  heart rate: 99003, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 7, 1 hour |  | 74
  heart rate: 99003, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 7, 4 hour |  | 73
  heart rate: 99003, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  heart rate: 99003, Day 7, 8 hour |  | 73
  heart rate: 99002, Day 1, pre-dose: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 1, pre-dose | 58 |
  heart rate: 99002, Day 1, 1 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 1, 1 hour | 62 |
  heart rate: 99002, Day 1, 4 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 1, 4 hour | 64 |
  heart rate: 99002, Day 1, 8 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 1, 8 hour | 73 |
  heart rate: 99002, Day 7, pre-dose: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 7, pre-dose | 68 |
  heart rate: 99002, Day 7, 1 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 7, 1 hour | 72 |
  heart rate: 99002, Day 7, 4 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 7, 4 hour | 67 |
  heart rate: 99002, Day 7, 8 hour: number analyzed (Participants) | 1 | 0
  heart rate: 99002, Day 7, 8 hour | 81 |

5. Secondary Outcome: Changes From Baseline to After Treatment in Faecal Calprotectin Levels
Description: Stool sample was collected from 1-hour post dose until 8 hours post dose for faecal calprotectin measures. It was not possible to draw any meaningful conclusions from the very limited data available. Data has been presented for the 3 participants (99001, 99002 and 99003) since the analysis was not done. Baseline was Day -1.
Time Frame: Day -1 and pre-dose and 8 hour post-dose on Day 1 and 7
Population: All subjects population.
Measure: Number; unit: milligram per litre (mg/L)
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
milligram per litre (mg/L)
  99002, Day1 pre-dose: number analyzed (Participants) | 1 | 0
  99002, Day1 pre-dose | 350.86 |
  99002, Day1 post dose (8 hour): number analyzed (Participants) | 1 | 0
  99002, Day1 post dose (8 hour) | 164.54 |
  99002, Day 7 pre-dose: number analyzed (Participants) | 1 | 0
  99002, Day 7 pre-dose | 430.30 |
  99002, Day 7 post dose (8 hour): number analyzed (Participants) | 1 | 0
  99002, Day 7 post dose (8 hour) | 524.90 |
  99003, Day1 pre-dose: number analyzed (Participants) | 0 | 1
  99003, Day1 pre-dose |  | 314.21
  99003, Day1 post dose (8 hour): number analyzed (Participants) | 0 | 1
  99003, Day1 post dose (8 hour) |  | 458.32
  99003, Day 7 pre-dose: number analyzed (Participants) | 0 | 1
  99003, Day 7 pre-dose |  | 306.15
  99001, Day1 pre-dose: number analyzed (Participants) | 0 | 1
  99001, Day1 pre-dose |  | 85.43
  99001, Day1 post dose (8 hour): number analyzed (Participants) | 0 | 1
  99001, Day1 post dose (8 hour) |  | 194.97
  99001, Day 7 pre-dose: number analyzed (Participants) | 0 | 1
  99001, Day 7 pre-dose |  | 134.04

6. Secondary Outcome: Amount of Medicine in Blood
Description: Blood samples were collected at 1, 2.25, 4, 8 hour on Day 1 and 7 for the analysis of amount of medicine in blood. It was not possible to draw any meaningful conclusions from the very limited data available. Data has been presented for the 3 participants (99001, 99002 and 99003) since the analysis was not done.
Time Frame: At 1, 2.25, 4, 8 hour on Day 1 and 7
Population: All subjects population.
Measure: Number; unit: nanogram per hour (ng/hr)
Arm/Group | SB656933 20 mg | SB656933 100 mg
Number analyzed (Participants) | 1 | 2
nanogram per hour (ng/hr)
  99001, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  99001, Day 1, 1 hour |  | 2831.20
  99001, Day 1, 2.25 hour: number analyzed (Participants) | 0 | 1
  99001, Day 1, 2.25 hour |  | 4293.70
  99001, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  99001, Day 1, 4 hour |  | 4107.40
  99001, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  99001, Day 1, 8 hour |  | 1234.80
  99001, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  99001, Day 7, 1 hour |  | 2893.90
  99001, Day 7, 2.25 hour: number analyzed (Participants) | 0 | 1
  99001, Day 7, 2.25 hour |  | 4238.70
  99001, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  99001, Day 7, 4 hour |  | 2722.40
  99001, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  99001, Day 7, 8 hour |  | 2005.00
  99003, Day 1, 1 hour: number analyzed (Participants) | 0 | 1
  99003, Day 1, 1 hour |  | 1076.80
  99003, Day 1, 2.25 hour: number analyzed (Participants) | 0 | 1
  99003, Day 1, 2.25 hour |  | 2606.90
  99003, Day 1, 4 hour: number analyzed (Participants) | 0 | 1
  99003, Day 1, 4 hour |  | 5192.70
  99003, Day 1, 8 hour: number analyzed (Participants) | 0 | 1
  99003, Day 1, 8 hour |  | 1288.50
  99003, Day 7, 1 hour: number analyzed (Participants) | 0 | 1
  99003, Day 7, 1 hour |  | 985.20
  99003, Day 7, 2.25 hour: number analyzed (Participants) | 0 | 1
  99003, Day 7, 2.25 hour |  | 1993.30
  99003, Day 7, 4 hour: number analyzed (Participants) | 0 | 1
  99003, Day 7, 4 hour |  | 3912.20
  99003, Day 7, 8 hour: number analyzed (Participants) | 0 | 1
  99003, Day 7, 8 hour |  | 1164.30
  99002, Day 1, 1 hour: number analyzed (Participants) | 1 | 0
  99002, Day 1, 1 hour | 438.30 |
  99002, Day 1, 2.25 hour: number analyzed (Participants) | 1 | 0
  99002, Day 1, 2.25 hour | 961.80 |
  99002, Day 1, 4 hour: number analyzed (Participants) | 1 | 0
  99002, Day 1, 4 hour | 562.30 |
  99002, Day 1, 8 hour: number analyzed (Participants) | 1 | 0
  99002, Day 1, 8 hour | 153.30 |
  99002, Day 7, 1 hour: number analyzed (Participants) | 1 | 0
  99002, Day 7, 1 hour | 616.10 |
  99002, Day 7, 2.25 hour: number analyzed (Participants) | 1 | 0
  99002, Day 7, 2.25 hour | 715.40 |
  99002, Day 7, 4 hour: number analyzed (Participants) | 1 | 0
  99002, Day 7, 4 hour | 944.20 |
  99002, Day 7, 8 hour: number analyzed (Participants) | 1 | 0
  99002, Day 7, 8 hour | 286.70 |

ADVERSE EVENTS:
Time Frame: Data for AE was collected up to follow-up (Visit 5) 7 to 10 days after last dose.
Description: The 'All Subjects population' was defined as all participants who received at least one dose of study medication. This population was used for the reporting of AEs.
Arm/Group | SB656933 20 mg | SB656933 100 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB656933 20 mg (N=1) | SB656933 100 mg (N=2)
Sensation of brick in stomach (Gastrointestinal disorders) | 0 | 1
herpes simplex (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was early terminated on 17 February 2010 because investigational drug and further that the duration of treatment (7 days) was unlikely to provide any clinical benefit to participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.